CLINICAL TRIAL: NCT05668143
Title: The Effect of Intraoperative Virtual Reality Application on the Level of Anxiety and Vital Findings in Patients Who Will Have Total Knee Replacement Surgery: A Randomized Controlled Study
Brief Title: Effect of Intraoperative Virtual Reality on Anxiety and Vital Findings in Patients Total Knee Replacement Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bucak State Hospital (Other Government)
Responsible Party: Principal Investigator, Yusuf Beşirik, Principal Investigator, Bucak State Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2022/008
Record Dates: First submitted 2022-12-09; First posted 2022-12-29 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Total Knee Replacement Surgery; Virtual Reality
Keywords: Intraoperative; Virtual Reality; Anxiety; Vital Findings; Patients; Total Knee Replacement Surgery
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The patients will be divided into two as the experimental and control group.The study will be conducted as a randomized controlled trial. Patients in the experimental group will be informed about the using virtual reality glasses during total knee replacement surgery.
Who Masked: Outcomes Assessor
Masking Description: Single Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): During the surgery, patients will be shown nature and landscape images with virtual reality glasses.
  Interventions: Behavioral: Virtual reality
- Control group (No Intervention): The control group will receive standard procedure without any intervention.

INTERVENTIONS:
Behavioral: Virtual reality — The Patient Information Form and the State Anxiety Scale will be administered to the patients just before the surgery. The researcher will measure the patient's respiratory, blood pressure, pulse and oxygen saturation values on the monitor just before the start of the operation and every 15 minutes after the operation, and the vital signs will be recorded in the follow-up form. Virtual reality glasses will be put on the patient immediately after anesthesia is given to the patient by the anesthesiologist. Glasses will be worn during the total knee replacement surgery. Total knee replacement surgery takes an average of 60 minutes. During the surgery, patients will be shown nature and landscape images with virtual reality glasses. Virtual reality glasses will be removed immediately after the operation and the State Anxiety Scale and vital signs follow-up form will be applied before the patient is sent to the service from the operating room.
  Arms: Experimental group

SUMMARY:
Although total knee replacement surgery improves the quality of life of the patients, a significant reduction in knee pain and normalization of the knee joint, the awareness of the surrounding events is a major concern for the patients and negatively affects their vital signs, since most of the patients are awake during the surgery. When the literature is examined, there are no pharmacological methods to reduce anxiety.

When distraction techniques are used, patients' anxiety levels are significantly reduced, vital signs are normalized, patient satisfaction is increased and pain is relieved.

It has been emphasized that there is a successful method in reducing One of the distraction techniques is the application of virtual reality. This study will be carried out in a randomized controlled experimental design to determine the effect of virtual reality application during surgery on patients who will undergo total knee replacement surgery, on the anxiety level and vital signs of the patients.

DETAILED DESCRIPTION:
The aim of this study is to determine the effect of virtual reality application on patients' anxiety level and vital signs during surgery for patients who will undergo total knee replacement surgery.

It will consist of patients over the age of 18 who will have total knee replacement surgery, which will be carried out in the Operating Room Unit. Patients meeting the sample selection criteria were randomized into experimental and control groups.

will be divided into two groups. Virtual reality glasses will be applied to the experimental group. In the collection of data; "Patient Information Form", "State Anxiety Inventory Scale" and "Vital Signs Follow-up Form" will be used.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily agreed to participate in the research
* Being 18 years or older
* Being able to read and write Turkish
* No vision and hearing problems
* Not using glasses
* Absence of any psychiatric, cognitive or neurological disease

Exclusion Criteria:

* Patients with visual or hearing impairment
* Patients receiving general anesthesia
* Those who have previously had total knee replacement surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-12-30 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
State Anxiety Scale | 10 minute
  State Anxiety Scale mean scores of the patients in the intervention and control groups will be compared before and after surgery. A minimum of 20 and a maximum of 80 points can be obtained from the scale. If the scale score approaches 80, it indicates high anxiety.
Respiratory Rate | 15 minute
  Just before the start of the operation and every 15 minutes after the operation, the patient's respiratory rate values will be measured on the monitor and the respiratory rate will be recorded in the follow-up form.
Blood Pressure (both systolic and diastolic blood pressure) | 15 minute
  Just before the start of the operation and every 15 minutes after the operation, the patient's blood pressure (both systolic and diastolic blood pressure) values will be measured on the monitor and the blood pressure (both systolic and diastolic blood pressure) will be recorded in the follow-up form.
Pulse | 15 minute
  Just before the start of the operation and every 15 minutes after the operation, the patient's pulse values will be measured on the monitor and the pulse will be recorded in the follow-up form.
Saturation Value | 15 minute
  Just before the start of the operation and every 15 minutes after the operation, the patient's saturation value will be measured on the monitor and the saturation will be recorded in the follow-up form.

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Beşirik, MScN student, Principal Investigator — Bucak State Hospital; Serap Sayar, PhD, Study Director — KTO Karatay University
Locations (1):
- Bucak State Hospital, Burdur, Turkey (Türkiye)